CLINICAL TRIAL: NCT03636867
Title: Prospective Evaluation of Laboratory, Cellular and Molecular Determinants of Clinical Success of the Treatment in Diabetic Patients With Critical Limb Ischemia (ECAD-CLI) Study
Brief Title: Laboratory, Cellular and Molecular Determinants of Clinical Success in Diabetic Patients With Critical Limb Ischemia
Acronym: ECAD-CLI
Status: Completed | Type: Observational
Sponsor: Maria Cecilia Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 5510/2018
Record Dates: First submitted 2018-08-13; First posted 2018-08-17 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus; Critical Limb Ischemia; Critical Lower Limb Ischemia; Diabetic Foot
MeSH Terms: conditions — Diabetes Mellitus; Chronic Limb-Threatening Ischemia; Diabetic Foot | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — for each patient, according clinical presentation and type of intervention, the Authors will collect: i) blood sample for DNA extraction, RNA extraction and serum collection; plaque from patients undergoing endoarterectomy, tissue removed from foot ulcers requiring debridement or surgical manipulation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- data and specimen collection: consecutive diabetic patients admitted to Maria Cecilia Hospital for critical limb ischemia
  Interventions: Other: data and specimen collection

INTERVENTIONS:
Other: data and specimen collection — to identify laboratory, cellular and molecular determinants of clinical success after treatment, several clinical information and specimens will be collected by Authors from each patient

SUMMARY:
The ECAD-CLI is an investigator-driven, prospective, single-center study. The aim of the study is to prospectively collect clinical, laboratory, angiographic, cellular and molecular variables related to prognosis and outcome in patients with diabetes mellitus and critical limb ischemia.

DETAILED DESCRIPTION:
All consecutive patients admitted to Maria Cecilia Hospital will be enrolled in the ECAD-CLI study. According to interventional management of the patient the following data and samples will be prospectively collected and related to outcome:

* medical history, cardiovascular risk factors, clinical presentation
* information related to angiography of peripheral arteries. An independent core-lab will review angiographies to assess extent and severity of peripheral artery disease
* information related to medical treatment, including antithrombotic agents, antimicrobics and any treatment to permit wound healing
* blood sample to obtain DNA, RNA and serum
* patient undergoing surgery and/or debridement for wound/ulcer due to diabetic foot disease will receive biopsy for specimen collection
* atherosclerotic plaque sample in patients undergoing atherectomy for the treatment of the peripheral artery disease All clinical variables and information obtained from blood/tissue samples will be related to outcome.

Any adverse events will be judged by an independent blinded committee.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of diabetes mellitus in treatment with oral agents and/or insulin
* diagnosis of critical limb ischemia requiring medical and/or interventional treatment

Exclusion Criteria:

* dialysis
* diagnosis or suspicion of malignancy
* life expectancy <1 year
* inability to guarantee clinical follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with diabetes mellitus and critical limb ischemia admitted to hospital for medical/interventional management of the disease
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Incidence of amputation | 1-year
  Occurrence of major or minor amputation

SECONDARY OUTCOMES:
Wound healing | 1-year
  occurrence of wound healing
Change in WIfI class | 1-year
  The Wound, Ischemia and Foot Infection is the most used classification for patients with diabetic foot disease. The classification ranges from 0 to 9. The scale includes 3 items: wound extension, presence and severity of ischemia, presence and severity of ischemia. Each item ranges from 0 to 3 points.
Change in Rutherford class | 1-year
  The Rutherford classification is the most used scale to stratify patients with peripheral artery disease. The classification ranges from class I to class VI. Patients with critical limb ischemia show a class from IV to VI. The Rutherford class will be assessed in all patients at baseline and 1-year after to estimate the presence or not of improvement
Incidence of revascularization of peripheral arteries | 1-year
  any procedure (percutaneous or surgical) of revascularization of peripheral arteries

OTHER OUTCOMES:
Incidence of major cardio and cerebrovascular adverse events (MACCE) | 1-year
  cumulative occurrence of all-cause death, myocardial infarction, cerebrovascular accident

CONTACTS AND LOCATIONS:
Overall Officials: Luca Dalla Paola, MD, Principal Investigator — Maria Cecilia Hospital; Gianluca Campo, MD, Principal Investigator — Università degli Studi di Ferrara
Locations (1):
- Maria Cecilia Hospital, Cotignola, Ravenna, Italy

IPD SHARING:
Plan to Share IPD: Undecided